CLINICAL TRIAL: NCT01206348
Title: A Phase IV, Open-Label Study Evaluating the Use of Solodyn (Minocycline HCL Extended-Release Tablets), Ziana, and Triaz Foaming Cloths as Combination Acne Therapy Prior to Treatment With Isotretinoin
Brief Title: Combination Treatment for Moderate to Severe Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medicis Global Service Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-0104-28
Record Dates: First submitted 2010-09-17; First posted 2010-09-21 (Estimated); Last update posted 2011-11-30 (Estimated); Status verified 2011-11

CONDITIONS: Acne
Keywords: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Minocycline; Clindamycin; Tretinoin; Benzoyl Peroxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label Combination (Experimental): Solodyn, Ziana, Triaz FC
  Interventions: Drug: Minocycline, Clindamycin, Tretinoin, Benzoyl Peroxide

INTERVENTIONS:
Drug: Minocycline, Clindamycin, Tretinoin, Benzoyl Peroxide — Solodyn 1 tablet, Q day Ziana Gel, topical Q am Triaz FC, topical Q night

SUMMARY:
To determine if a combination of three currently approved acne products are safe and effective for the treatment of moderate to severe acne

DETAILED DESCRIPTION:
A Phase IV, Open-Label Study Evaluating the treatment for Combination Acne Therapy.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe acne, IGA = 3 or 4 (Investigator Global Assessment)

Exclusion Criteria:

* pregnancy and allergies

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2010-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients showing improvement from Baseline and Week 12 | Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Mary Sanstead, BSN, CCRP, Study Chair — Medicis Global Service Corporation
Locations (10):
- United States (10):
  - Birmingham, Alabama
  - Santa Monica, California
  - Hockessin, Delaware
  - Chestnut Hill, Massachusetts
  - Detroit, Michigan
  - Henderson, Nevada
  - High Point, North Carolina
  - Hershey, Pennsylvania
  - Nashville, Tennessee
  - Salt Lake City, Utah